CLINICAL TRIAL: NCT04390412
Title: Assessment of Adding Low Dose Pulmonary Radiotherapy to the National Protocol of COVID-19 Management: A Pilot Trial
Brief Title: Low Dose Radiotherapy in COVID-19 Pneumonia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23568; IRCT20200509047366N1 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-07

CONDITIONS: COVID; SARS (Severe Acute Respiratory Syndrome)
Keywords: Low Dose Lung Radiotherapy; COVID-19; anti-inflammatory
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose Radiotherapy (Experimental): 0.5 Gy radiation to both lungs in an AP/PA fashion
  Interventions: Radiation: Low Dose Radiotherapy

INTERVENTIONS:
Radiation: Low Dose Radiotherapy — 0.5 Gy radiation to both lungs in an AP/PA treatment plan

SUMMARY:
Moderate to severe cases of SARS-associated ARDS based on inclusion/ exclusion criteria and the decision made in multi- disciplinary team are treated with 0.5 Gy whole lung radiation.

DETAILED DESCRIPTION:
SARS-associated ARDS (acute respiratory distress syndrome) is the most fatal outcome of COVID-19 systemic infection. To overcome the uncontrolled inflammation leading to ARDS and respiratory failure, several drugs have been investigated in this situation with the most promising results coming from anti-inflammatory agents that directly or indirectly inhibit IL-6 and its counterparts of inflammation.

Low dose radiation, as opposed to high dose, has documented anti-inflammatory effects that are exercised through various mechanisms including decrease in pro-inflammatory cytokines such as IL-6.

In this pilot clinical trial, the patients are carefully selected according to inclusion /exclusion criteria and the clinical judgement of the multi- disciplinary team.Their diagnostic CT scan will be used to plan an AP/ PA radiotherapy treatment to both lungs and the set-up positioning information is obtained from anatomical landmarks. The patient will be referred for a fraction of 0.5 Gy to both lungs and for the next 28 days the clinical para-clinical and radiologic variables of disease severity will be monitored closely. Should the patient's clinical course indicate and the multi- disciplinary team approves, they may be subjected to another fraction of 0.5 Gy to a maximum of 1 Gy in two fractions at least 72 hours apart. All the patients will also receive the standard national protocol of COVID-19 management.

A total of 5 patients will be enrolled in the RT arm, providing favourable results seen in the first set of patients, the team will decide on recruiting a larger number for a phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 diagnosis ( PCR or serologic or radiographic)
* Presence of pulmonary involvement ( defined by P/F ratio or NIV need)
* Less than 3 days since the onset of ARDS
* Age > 60 years
* ↑ IL-6 ( if available)
* ↑ CRP

Exclusion Criteria:

* Lack of informed consent
* Inability to transfer to the radiation unit
* Hemodynamic instability
* Septic shock and organ dysfunction
* Severe ARDS P/F ratio ≤ 100 mmHg
* History of cardiac failure
* Contraindications to radiation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline blood oxygenation | 28 days
  O2 saturation
Number of Hospital stay days | 28 days
  Total days the patient is admitted to hospital
Number of ICU stay days | 28 days
  Total days the patient is admitted to ICU
Number of intubation events | 28 days
  Total number of intubations performed after the treatment

SECONDARY OUTCOMES:
WBC | 28 days
  Changes in WBC count if base-line is abnormal
Platelets | 28 days
  Changes in Platelets count if base-line is abnormal
CRP | Day 1
  Changes in CRP serum level
CRP | Day 2
  Changes in CRP serum level
CRP | Day 3
  Changes in CRP serum level
CRP | Day 4
  Changes in CRP serum level
CRP | Day 5
  Changes in CRP serum level
IL-6 | Day 1
  Changes in IL-6 serum level
IL-6 | Day 2
  Changes in IL-6 serum level
IL-6 | Day 3
  Changes in IL-6 serum level
IL-6 | Day 4
  Changes in IL-6 serum level
IL-6 | Day 5
  Changes in IL-6 serum level

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Ameri, Prof., Study Chair — Shahid Beheshti University of Medical Sciences; Nazanin Rahnama, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Imam Hossein Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after the completion of study to other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion of trial for one year.
Access Criteria: Verified researchers

REFERENCES:
- [Background] Calabrese EJ, Dhawan G. How radiotherapy was historically used to treat pneumonia: could it be useful today? Yale J Biol Med. 2013 Dec 13;86(4):555-70. PMID 24348219
- [Background] Large M, Hehlgans S, Reichert S, Gaipl US, Fournier C, Rodel C, Weiss C, Rodel F. Study of the anti-inflammatory effects of low-dose radiation: The contribution of biphasic regulation of the antioxidative system in endothelial cells. Strahlenther Onkol. 2015 Sep;191(9):742-9. doi: 10.1007/s00066-015-0848-9. Epub 2015 Jun 8. PMID 26051282
- [Background] Clayton B. Hess, MD, MPH, and Mohammad K. Khan, MD, PhD, "Low dose chest radiation for COVID-19 patients" Winship Emory News post, April 27, 2020
- [Background] Kirkby C, Mackenzie M. Is low dose radiation therapy a potential treatment for COVID-19 pneumonia? Radiother Oncol. 2020 Jun;147:221. doi: 10.1016/j.radonc.2020.04.004. Epub 2020 Apr 6. No abstract available. PMID 32342871
- [Background] Kefayat A, Ghahremani F. Low dose radiation therapy for COVID-19 pneumonia: A double-edged sword. Radiother Oncol. 2020 Jun;147:224-225. doi: 10.1016/j.radonc.2020.04.026. Epub 2020 Apr 20. No abstract available. PMID 32342874
- [Background] Stefano M Magrini, Prof et al. COVID-19 Pneumonitis Low Dose Lung Radiotherapy (COLOR-19). ClinicalTrials.gov Identifier: NCT04377477